CLINICAL TRIAL: NCT05942573
Title: SCAFIGC：Continuation of Serplulimab Plus Chemotherapy After First Progression in Advanced Gastric or Gastro-oesophageal Junction Adenocarcinoma: an Open-label, Randomised Phase II Trial
Brief Title: Continuation of Serplulimab Plus Chemotherapy After First Progression in Advanced Gastric or Gastro-oesophageal Junction Adenocarcinoma: an Open-label, Randomised Phase II Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCAFIGC
Record Dates: First submitted 2023-04-17; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2022-10

CONDITIONS: Gastric Cancer (GC) Gastroesophageal Junction Cancer (GEJ)
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Serplulimab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- continuation of Serplulimab plus chemotherapy after first progression (Experimental): Serplulimab+Paclitaxel+Apatinib
  Paclitaxel±Ramucirumab
  Interventions: Drug: Serplulimab+Paclitaxel+Apatinib; Drug: Paclitaxel±Ramucirumab

INTERVENTIONS:
Drug: Serplulimab+Paclitaxel+Apatinib — Immunotherapy+chemotherapy
  Other Names: A:Drug:Serplulimab+paclitaxel+Apatinib
Drug: Paclitaxel±Ramucirumab — chemotherapy±Targeted therapy
  Other Names: B:Drug:paclitaxel±Ramucirumab

SUMMARY:
This study is conducted in patients with advanced metastatic gastric cancer including gastroesophageal junction cancer(patients with HER2 negative and PD-L1 CPS≥5).Patiens will recevie Serplulimab plus chemotherapy ((oxaliplatin+capecitabine) as first-line treatment. After PD，patients will randomly 2：1 assigned to treatment：one group will receive Serpluimab with Paclitaxel,Apatinib；another group will receive Paclitaxel with or without Ramucirumab.All of eligible patients will receive study drug treatment until loss of clinical benefit, unacceptable toxicity, death, withdrawal of informed consent

DETAILED DESCRIPTION:
stage one ：Serplulimab 3mg/kg,d1,q2w or 4.5mg/kg,d1,q3w+oxaliplatin130mg/m2 iv.gtt d1+capecitabine 1000mg/m2 p.o.b.i.d d1~d14,q3w

stage two:Serplulimab 3mg/kg,d1,q2w or 4.5mg/kg,d1,q3w+Apatinib 250mg/qd+Paclitaxel 135~175mg/m2 iv.gtt,d1,q3w

Paclitaxel 135~175mg/m2 iv.gtt,d1,q3w±Ramucirumab 8mg/kg,d1,q2w

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in this clinical study; completely understand and know this study as well as sign the informed consent form (ICF); be willing to follow and be able to complete all study procedures;
2. Age ≥ 18 years and ≤ 75 years when ICF is signed;
3. Unresectable locally advanced, or metastatic gastric cancer including gastroesophageal junction cancer, and histopathologically confirmed diagnosis of adenocarcinoma;
4. never received systemic anti-tumor drug therapy before；
5. HER2 negative and PD-L1 CPS≥5;
6. Measurable lesion according to RECIST v1.1 by IRRC;
7. ECOG score 0-1;

Exclusion Criteria:

1. Has other active malignancies within 5 years before the first administration of the study drug;
2. Plan to or have previously received organ or bone marrow transplantation;
3. Uncontrollable pleural effusion, pericardial effusion or ascites requiring repeated drainage;
4. Have received any research drugs within 14 days before the first use of the study drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2022-12-24 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
6-month PFS% | The Percent of patinets after first progression until disease progression in 6 months
  Progression-free survival by IRRC assessment per RECIST 1.1

SECONDARY OUTCOMES:
OS | From the date of first dose unitl the date of death from any cause，assessed up to 2 years ]
  Overall survival
PFS2 | From date of randomization until the date of second-line treatment progression or date of death from any cause, whichever came first
  Progression-free survival by IRRC assessment per RECIST 1.1
PFS1 | From date of randomization until the date of first documented progressionor date of death from any cause, whichever came first
  Progression-free survival by IRRC assessment per RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No